CLINICAL TRIAL: NCT05285852
Title: The Effects of Triggering Points Dry Needling on Sternocleidomastoid Muscle for Pain and Disability in Migraine
Brief Title: Effects Of Dry Needling On Sternocleidomastoid Muscle For Pain And Disability In Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-FSD-00258
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Migraine
Keywords: Dry Needling; Sternocleidomastoid Muscle; Pain; Disability; Randomized Control Trial; Migraine
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): For application of the Dry Needling the individual should be in the supine position. To facilitate the approach and adhesion of the Sternocleidomastoid Muscle, the person's neck is placed ipsilaterally in the slightly lateral flexed position. Consequently, the therapist identified the active Trigger Points in the Sternocleidomastoid Muscle and cleansed the surface using an antiseptic solution. Using the insertion pipe, the dry needle inserted into the muscle. For the separation of neurovascular structure from muscle belly the needle is carried out in an anterior-posterior direction. A compression of 90 secs with a cotton swab will be applied at the needling site immediately after removing the needle to reduce the intensity and duration of pain. The variables will then be measured immediately following the processing session. Six sessions of Dry Needling will be applied to each patient and there will be a gap of at least 48 hours between each session.
  Interventions: Other: Dry Needling
- Placebo Dry Needling (Placebo Comparator): Following identification of the trigger point in the muscle, the surface would be cleaned with an antiseptic solution. For placebo Dry Needling, which only causes a pricking sensation, a blunt needle will be applied to the trigger points without penetrating the skin after application of a certain pressure to the skin. The protocol will be applied six times, with a two-day pause between treatments. Like the intervention group, the variables will be measured immediately after the processing session.
  Interventions: Other: Placebo Dry Needling

INTERVENTIONS:
Other: Dry Needling — Dry needling technique is maneuvered by different skilled health practitioners aiming to reduce central sensitization, i.e., the hypersensitivity to pain of the central nervous system. It is also apprehended to reduce the local and referred pain, and improve the muscle activation patterns leading to improved range of motion.
  Arms: Dry Needling
Other: Placebo Dry Needling — Placebo Dry Needling only causes a pricking sensation
  Arms: Placebo Dry Needling

SUMMARY:
To determine the effects, sequel of dry needling in migraine by resolving MTrPs in sternocleidomastoid muscle.

To determine the possession of dry needling technique to mitigate the frequency, intensity and duration of headache.

To determine the effectiveness of dry needling in the disability hindrance in migraine patients.

DETAILED DESCRIPTION:
This is a randomized control study of 60 volunteers with migraine induced by myofacial triggers in sternocleidomastoid muscle. The migraine will be diagnosed by the neurologist and for the evaluation of trigger points and muscle thickness ultrasound will be done. After the diagnostic procedure and complete history evaluation from the selected population 30 subjects will be subjected to dry needling group and 30 others will be kept in the placebo group. All the participants will receive six sessions at the myofascial trigger point area there should be the gap of at least 48 hours between two sessions. As for the assessment details, such as the frequency, intensity and duration of the headaches; the consumption of drugs; the thickness of SCM muscles; the pain pressure threshold and the cervical range motions will be recorded before, immediately following the response, and at the 1-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Submitted with a headache diagnosis by a neurologist.
* Presence of active Trigger points in the Sternocleidomastoid muscle reproducing the symptoms of migraine.
* Active trigger points will be identified if "there is muscle sensitivity that has been activated by pressure and reproduces the patient's referred pain and headache."
* A jump sign the characteristic behavioral response to compression on a trigger point, will be produced.

Exclusion Criteria:

* background of neck trauma
* cervical radiculopathy
* History of head/shoulder surgery
* Diagnosis of other unusual headaches/migraines
* Phobia of pricking
* pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12th Week
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Bubble Inclinometer | 12th Week
  Bubble Inclinometer is a simple to use device for measuring range of motion in patients. The inclinometer can be used to measure range of motion in the neck, the hip, the elbow, the knee, the shoulder, the spine, the ankle, the wrist, and the Metacarpophalangeal joint.
Sternocleidomastoid muscle Ultrasonography | 12th Week
  An ultrasonograph scan uses high-frequency sound waves to make an image of a person's internal body structures

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No